CLINICAL TRIAL: NCT03746301
Title: Xarelto® on Prevention of Stroke and Non-Central Nervous Systemic (CNS) Embolism in Renally Impaired Korean Patients With Non-valvular Atrial Fibrillation (NVAF)
Brief Title: Xarelto on Prevention of Stroke and Non-Central Nervous Systemic Embolism in Renally Impaired Korean Patients With Non-valvular Atrial Fibrillation
Acronym: XARENAL
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Collaborators: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: 20286
Record Dates: First submitted 2018-11-16; First posted 2018-11-19 (Actual); Last update posted 2022-12-08 (Actual); Status verified 2022-12

CONDITIONS: Non-valvular Atrial Fibrillation (NVAF)
Keywords: Non-valvular Atrial fibrillation (NVAF), Stroke; Non-Central Nervous Systemic (CNS) embolism
MeSH Terms: conditions — Stroke; Embolism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Treatment: Patients will be followed according to routine medical practice and the frequency of visits and procedures will be performed under routine conditions.
  Interventions: Drug: Rivaroxaban(Xarelto,BAY 59-7939)

INTERVENTIONS:
Drug: Rivaroxaban(Xarelto,BAY 59-7939) — 10mg, 15mg and 20 mg film-coated tablets

SUMMARY:
The purpose of the study is to evaluate the safety and effectiveness of Xarelto in renally impaired patients with NVAF under routine practice conditions. The information collected in the XARENAL study will help to understand how renally impared patients with NVAF are treated in the real-world setting and what the outcome for the patients is under those conditions.

ELIGIBILITY:
Inclusion Criteria:

* Female and male patients ≥ 19 years of age
* Diagnosis of NVAF
* Patients for whom the decision to initiate treatment with rivaroxaban has already been made as per physician's routine treatment practice
* Previous documented creatinine clearance rate of 15-49mL/min within 6 months before enrollment
* Written informed consent of the patient

Exclusion Criteria:

* Contraindications for rivaroxaban according to the current Korean market authorization and Summary of Product Characteristics (SmPC).
* Patients participating in an investigational program with interventions outside of routine clinical practice.
* Planned treatment with other anticoagulants.
* Expected renal-replacement therapy within the next 3 months

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with NVAF who have moderate (creatinine clearance 30 - 49 ml/min) or severe (creatinine clearance 15 - 29 ml/min) renal impairment, requiring rivaroxaban for the prevention of stroke or non-CNS systemic embolism. Patients must also meet all the eligibility criteria for the study.
Sampling Method: Non-Probability Sample
Enrollment: 924 (Actual)
Dates: Start 2018-12-03 (Actual); Primary Completion 2021-07-28 (Actual); Study Completion 2021-12-15 (Actual)

PRIMARY OUTCOMES:
Incidence proportion of major bleeding | Up to 12 months
  Incidence proportion of major bleeding events collects as serious or non-serious AEs and defined as overt bleeding associated with:
  * a fall in haemoglobin of ≥2 g/dL, or
  * a transfusion of ≥2 units of packed red blood cells or whole blood, or
  * occurrence at a critical site (intracranial, intra-spinal, intraocular, pericardial, intra articular, intra muscular with compartment syndrome, retroperitoneal), or
  * death.

SECONDARY OUTCOMES:
Occurrence of AEs and SAEs | Up to 12 months
Occurrence of all-cause mortality | Up to 12 months
Occurrence of Non-major bleeding | Up to 12 months
  Non-major bleeding events collected as SAEs or non-serious AEs and defined as all bleeding events that do not fall in the category of major bleeding.
Incidence proportion of Symptomatic thromboembolic events | Up to 12 months
  Symptomatic thromboembolic events collected as SAEs or non-serious AEs.
Days of rivaroxaban treatment | Up to 12 months
  Start of rivaroxaban therapy and, if applicable, stop of rivaroxaban therapy(in case of treatment discontinuation, switch, or interruption, the reason will be recorded)
The change in creatinine clearance from baseline | At month 3,6,9 and 12

CONTACTS AND LOCATIONS:
Locations (1):
- Many locations, Multiple Locations, South Korea

IPD SHARING:
Plan to Share IPD: No
Availability of this study's data will later be determined according to Bayer's commitment to the EFPIA/PhRMA "Principles for responsible clinical trial data sharing". This pertains to scope, timepoint and process of data access. As such, Bayer commits to sharing upon request from qualified researchers patient-level clinical trial data, study-level clinical trial data, and protocols from clinical trials in patients for medicines and indications approved in the US and EU as necessary for conducting legitimate research. This applies to data on new medicines and indications that have been approved by the EU and US regulatory agencies on or after January 01, 2014.
  Interested researchers can use www.vivli.org to request access to anonymized patient-level data and supporting documents from clinical studies to conduct research. Information on the Bayer criteria for listing studies and other relevant information is provided in the member section of the portal.

REFERENCES:
- [Derived] Oh IY, Lee CH, Choi EK, Lim HE, Oh YS, Choi JI, Ahn MS, Kim JY, Kim NH, Yoon N, Sandmann M, Choi KJ. A Real-World, Prospective, Observational Study of Rivaroxaban on Prevention of Stroke and Non-Central Nervous Systemic Embolism in Renally Impaired Korean Patients With Non-Valvular Atrial Fibrillation: XARENAL. Korean Circ J. 2025 Feb;55(2):121-131. doi: 10.4070/kcj.2024.0154. Epub 2024 Oct 23. PMID 39601397
- See also: Click here to find information for studies related to Bayer products. To find this study enter the ClinicalTrials.gov identifier (NCT) number or Bayer Study Identifier (ID) in the search field. — http://clinicaltrials.bayer.com/